CLINICAL TRIAL: NCT03874065
Title: Formation of a Precision Oncology Registry
Brief Title: Medical Data Collection in the Formation of Precision Oncology Registry
Status: Terminated | Type: Observational
Why Stopped: PI left institution
Sponsor: Wake Forest University Health Sciences (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Other Study IDs: IRB00054757; NCI-2019-01293 (Registry Identifier: Clinical Trial Reporting Program); P30CA012197 (NIH); CCCWFU 04218 (Other: Wake Forest Baptist Comprehensive Cancer Center)
Record Dates: First submitted 2019-03-08; First posted 2019-03-14 (Actual); Last update posted 2024-01-19 (Actual); Status verified 2024-01

CONDITIONS: Cancer
MeSH Terms: conditions — Neoplasms

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 2 Years
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: Medical Chart Review — Collection of data from participant's medical chart

SUMMARY:
In efforts to develop an aggregation point for patient clinical data and data related to DNA sequencing in the Comprehensive Cancer Center, this registry will be developed to provide a comprehensive data store. The goal of the registry will be to collect information on the Cancer Center population undergoing next generation DNA sequencing (NGS) on their tumors or liquid biopsies.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To capture characteristics of the patient population undergoing next generation deoxyribonucleic acid (DNA) sequencing of their tumor or liquid biopsy for more efficient clinical operations by collecting data on demographics, disease, and previous treatment.

II. To gather information on the number and type of patients that receive off label, standard, timeline or other experimental treatments based on the next generation sequencing (NGS) data.

III. To gather data regarding the patient population that may require financial assistance.

IV. To describe the patient population, in terms of demographic and clinical characteristics, who have consented to have their next generation sequencing data to be linked to their clinical records and used for future research.

V. To collect overall survival for those patients with next generation sequencing data.

VI. To collect outcomes and response to the standard, experimental and/or off label treatment.

OUTLINE: Participants undergo collection of medical data to be used in the formation of a precision oncology registry. Medical data is collected as long as patients are receiving treatment for cancer.

ELIGIBILITY:
Inclusion Criteria:

• All cancer patients at Wake Forest Baptist Comprehensive Cancer Center and its satellites who are having next generation DNA sequencing ordered/performed on their tumor biopsy or surgically resected tissue and/or blood samples.

Exclusion Criteria: Not applicable

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: The population of the registry will be comprised of Wake Forest Baptist Comprehensive Cancer Center cancer patients undergoing NGS from their tumor or liquid biopsy.
Sampling Method: Probability Sample
Enrollment: 2885 (Actual)
Dates: Start 2019-05-17 (Actual); Primary Completion 2024-01-11 (Actual); Study Completion 2024-01-11 (Actual)

PRIMARY OUTCOMES:
Data Collection of Demographics, Disease and Previous Treatment | Approximately 2 years
  To capture characteristics of the patient population undergoing next generation DNA sequencing of their tumor or liquid biopsy for more efficient clinical operations by collecting data on demographics, disease, and previous treatment.
Modes of Treatment for Patients | Approximately 2 years
  To gather information on the number and type of patients that receive off label, standard, timeline or other experimental treatments based on the NGS data.
Populations Requiring Financial Assistance | Approximately 2 years
  To gather data regarding the patient population that may require financial assistance
Demographics Collection to Assess Patient Population | Approximately 2 years
  To describe the patient population, in terms of demographic, who have consented to have their NGS data to be linked to their clinical records and used for future research
Clinical Characteristics of Disease | Approximately 2 years
  To describe the patient population, in terms clinical characteristics, who have consented to have their NGS data to be linked to their clinical records and used for future research
Overall Survival | Approximately 2 years
  To collect overall survival for those patients with NGS data
Outcome and Response to Different Forms of Treatment | Approximately 2 years
  To collect outcomes and response to the standard, experimental and/or off label treatment

CONTACTS AND LOCATIONS:
Overall Officials: Stefan Grant, MD, Principal Investigator — Wake Forest University Health Sciences
Locations (1):
- Wake Forest Baptist Comprehensive Cancer Center, Winston-Salem, North Carolina, United States

IPD SHARING:
Plan to Share IPD: No
No reference to any individual participant will appear in reports, presentations, or publications that may arise from the collection of this data. The data could be used for a research study. All data provided for research will be completely deidentified.